CLINICAL TRIAL: NCT00624546
Title: Effect of Antireflux Therapy on the Expression of Genes Known to be Important in Inflammation, Metaplasia and Neoplasia in Patients With GERD
Brief Title: Effect of Antireflux Therapy on the Expression of Genes in Patients With GERD
Status: Terminated | Type: Observational
Why Stopped: Expected recruitment numbers have not been achieved.
Sponsor: University of Rochester (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey H Peters, Professor and Chair of the Department of Surgery, University of Rochester
Other Study IDs: RSRB18199; rsrb18199
Record Dates: First submitted 2007-12-28; First posted 2008-02-27 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: GERD; Gastroesophageal Reflux
Keywords: GERD; gastroesophageal reflux; antireflux surgery; Barrett's; Esophagus; Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Esophageal mucosal biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: gerd patients
  Interventions: Drug: Prevacid Solutabs; Procedure: Antireflux surgery
- 2: non gerd controls

INTERVENTIONS:
Drug: Prevacid Solutabs — BID Prevacid Solutabs
  Groups: 1
Procedure: Antireflux surgery — Lap Nissen
  Groups: 1

SUMMARY:
Although the symptomatic and epithelial (histologic and endoscopic) response to antireflux therapy are well known and extensively studied, little is known of the genetic events occurring in response to proton pump inhibitor therapy. Preliminary data from our laboratory has shown, for example, that COX-2 expression is not only elevated in patients with gastroesophageal reflux disease but also can be correlated with pathologic esophageal acid exposure on 24 hour pH monitoring. Similar studies have suggested that antireflux surgery may normalize COX-2 gene expression. In contrast studies following ablation of dysplastic Barrett's epithelium have shown persistence of genetic changes associated with altered cellular function, despite the return of the histologic appearance to normal. Several key mediators of inflammation, metaplasia (Barrett's) and neoplasia have now been well characterized and shown to be important factors in the pathogenesis of esophageal injury. It is likely that successful antireflux therapy returns altered expression of these mediators toward normal although this hypothesis remains largely unexplored. The aim of this study is to investigate gene expression of key mediators of the spectrum of esophageal mucosal injury and the response to antireflux therapy.

Hypothesis: Antireflux therapy (proton pump inhibitor and surgical fundoplication) normalizes the expression of genes known to be involved in the pathogenesis of inflammation (esophagitis), metaplasia (Barrett esophagus) and neoplasia (adenocarcinoma).

DETAILED DESCRIPTION:
Aims: To determine the effects of antireflux therapy (pump inhibitor and surgical fundoplication) on gene expression of:

1. inflammation: IL-8, IFN-g, TNF-a.
2. intestinal metaplasia: CDX-1/2, MUC2 and Sonic hedgehog.
3. Neoplasia: Cox-2, VEGF, and EGFR.

ELIGIBILITY:
Inclusion Criteria:

For patients with GERD

* Patients referred for anti-reflux surgery
* On PPI therapy for at least 6 months
* Positive ambulatory pH monitoring (%time pH<4 > 4.7)
* Age greater than 18 years old.
* Both genders

For non-GERD controls

* Negative ambulatory pH monitoring OR
* Upper endoscopy performed for non-GERD symptoms.
* Age greater than 18 years old.
* Both genders

Exclusion Criteria:

* Prior foregut surgery
* Contra-indications for operation (poor clinical status, etc.)
* Contra-indications for endoscopy and biopsy (esophageal or gastric varices, therapeutic anticoagulation with Coumadin or Heparin, etc.)
* Unwillingness to participate in all of the follow-up studies
* Pregnancy
* Patients using medications that may interfere with PPIs pharmacokinetics (sucralfate, ketoconazole (Nizoral), ampicillin (Omnipen, Principen), digoxin (Lanoxin, Lanoxicaps), and iron (Feosol, Mol-Iron, Fergon, Femiron).
* Patients using medications that may interfere with gene expression (Immunosuppressants, Aspirin, NSAIDs, Corticosteroids).
* Patients with diseases that may interfere with gene expression (autoimmune diseases, diseases that course with immunosuppression).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects: (a) 20 patients with GERD and (b) 20 non-GERD controls.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
gene expression | before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Peters, Principal Investigator — University of Rochester
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States